CLINICAL TRIAL: NCT04309617
Title: Provider Referral Patterns Following Nephrectomy in High-Risk Locoregional Renal Cell Carcinoma
Brief Title: Retrospective Study on Referral Patterns for High Risk Patients Post Nephrectomy
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181230
Record Dates: First submitted 2020-03-13; First posted 2020-03-16 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with Renal Cell Carcinoma(RCC): Patients diagnosed with RCC who received a nephrectomy between 01Apr2014 and 31Mar2019
  Interventions: Procedure: nephrectomy

INTERVENTIONS:
Procedure: nephrectomy — Surgery performed within the study period

SUMMARY:
This study aims at estimating the proportion of patients diagnosed with locoregional renal cell carcinoma who are at high risk for recurrence following nephrectomy, describe referral patterns, and characterize treatment in this population. Outcomes including estimation of the incidence of recurrence and disease-free interval following nephrectomy will be reported overall and among the subgroup off patients receiving adjuvant systemic therapy with sunitinib following nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for data abstraction:

  * Diagnosed with locoregional RCC (no distant metastasis at the time of diagnosis)
  * Underwent a nephrectomy at Duke between 01 April 2014, and 31 December 2019 (final dates determined based on results from part 2 data collection)
  * Aged 18 years or older at nephrectomy

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who were diagnosed with locoregional RCC and underwent nephrectomy at Duke
Sampling Method: Non-Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Dzimitrowicz H, Esterberg E, Miles L, Zanotti G, Borham A, Harrison MR. Referral and adjuvant treatment patterns after nephrectomy in high-risk locoregional renal cell carcinoma. Cancer Med. 2021 Dec;10(24):8891-8898. doi: 10.1002/cam4.4407. Epub 2021 Nov 9. PMID 34751002
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical record data, for participants with locoregional renal cell carcinoma (RCC), who were recommended to go through nephrectomy at Duke from 01 April 2014 to 31 December 2019, were compiled retrospectively by Duke researchers via an institutional database.
Pre-assignment Details: Data collected were observed and evaluated in this study's duration of approximately 9 months.
Groups:
- All Participants: Eligible participants diagnosed with locoregional RCC who were recommended to go through nephrectomy at Duke from 01 April 2014 to 31 December 2019 were included and their data from medical records were evaluated and observed in the study.
Period: Overall Study
Arm/Group | All Participants
Started | 618
Modified High Risk of Recurrence | 136
Completed | 618
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved from medical records and studied.
Arm/Group | All Participants
Number analyzed (Participants) | 618
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (11.15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 417
  Female | 200
  Other | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 460
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 57
  Race: White | 103
  Race: Missing | 458
Time from RCC Diagnosis to Nephrectomy [Mean (Standard Deviation); unit: days] — Population: In this baseline measure, duration (in days) from time of RCC diagnosis to nephrectomy was reported. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this baseline measure.
  days
    number analyzed (Participants) | 616
    (all) | 5.03 (69.50)
Number of Participants Classified According to Tumor, Node, Metastasis (TNM) stage [Count of Participants; unit: Participants] — In this baseline measure, participants were classified according to their TNM stage. T = size and extent of the main tumor, N = number of nearby lymph nodes that have cancer and M = whether the cancer has metastasized. There are 4 TNM stages from 1 to 4, in which participants were distributed. Stage 1 to 3 refers to cancer is present; higher the stage larger the cancer tumor and more it has spread into nearby tissues. Stage 4 refers to the cancer has spread to distant parts of the body.
  Participants
    Stage 1 | 420
    Stage 2 | 65
    Stage 3 | 133
    Stage 4 | 0
Number of Participants Classified According to Tumor Fuhrman (Nuclear) Grade [Count of Participants; unit: Participants] — In this baseline measure, participants were classified according to Fuhrman (nuclear) grade. Grade 1= round or uniform nuclei; nucleoli not discernible or absent; Grade 2= slightly irregular nuclear contours; nucleoli visible at 400X (400 times its actual size); Grade 3= moderately to markedly irregular nuclear contours; nucleoli visible at 100X (100 times its actual size); Grade 4= multilobular nuclei or bizarre nuclei and large and prominent nucleoli. Population: Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 595
    Grade 1 | 71
    Grade 2 | 401
    Grade 3 | 95
    Grade 4 | 28
Number of Participants Classified According to Clear Cell Predominance [Count of Participants; unit: Participants] — In this baseline measure, participants were classified as "Yes" if they had a clear cell predominance or "No" if they did not had a clear cell predominance.
  Participants
    Yes | 457
    No | 161
Mean Tumor Size [Mean (Standard Deviation); unit: centimeter] — Population: In this baseline measure, mean tumor size of participants was reported. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this baseline measure.
  centimeter
    number analyzed (Participants) | 616
    (all) | 5.27 (3.39)
Number of Participants Classified According to Tumor Necrosis [Count of Participants; unit: Participants] — Population: In this baseline measure, participants were classified per presence or absence of tumor necrosis. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 614
    Present | 156
    Absent | 458
Number of Participants Classified According to Nephrectomy Year [Count of Participants; unit: Participants] — In this baseline measure, number of participants were classified according to year when they underwent nephrectomy.
  Participants
    2014 | 0
    2015 | 80
    2016 | 131
    2017 | 120
    2018 | 128
    2019 | 159
Number of Participants Classified According to Type of Nephrectomy [Count of Participants; unit: Participants] — In this baseline measure, number of participants according to type of nephrectomy they underwent (full or partial) were reported.
  Participants
    Full | 295
    Partial | 323
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG scale: 0=fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about >50% of waking hours; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair. Population: Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 269
    0 | 132
    1 | 129
    2 | 8
    3 | 0
    4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Follow-up Duration
Description: Follow- up time (in years) was duration between index date to the last entry in the medical record, death, or disease recurrence. The date of nephrectomy was considered as index date.
Time Frame: From index date to the last entry in the medical record, death, or disease recurrence, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and studied.
Measure: Median (Full Range); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 618
years | 1.07 [0.00 to 4.87]

2. Primary Outcome: Number of Participants Classified According to Follow-up Plan Determined at First Post-operative Visit
Description: In this outcome measure number of participants were classified according to their follow-up plan determined at first post-operative visit. Follow-up plans were as follows: 1) surveillance, 2) adjuvant systemic therapy (AST), 3) follow-up plan not recorded in the medical record and 4) other.
Time Frame: At first post-nephrectomy visit during approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and studied. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Eligible participants diagnosed with loco regional RCC who were recommended to go through nephrectomy at Duke from 01 April 2014 to 31 December 2019 were included and their data from medical records were evaluated and observed in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 552
Participants
  Surveillance | 519
  AST | 25
  Not Recorded | 5
  Other | 3

3. Primary Outcome: Number of Participants With Transfer of Care to a Non-Duke Provider
Description: In this outcome measure number of participants with transfer of care to a non-Duke provider were reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 536
Participants | 36

4. Primary Outcome: Number of Participants With no Documented Oncologic/RCC Related Care Referrals: Modified High Risk Sub-group
Description: Among number of participants who were followed up for any referral, those participants who had no documented oncologic/RCC related care referrals were recorded and reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: Post-nephrectomy approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here 'Overall Number of Participants Analyzed' signifies participants who were followed up for evaluation for any referral.
Measure: Count of Participants; unit: Participants
Groups:
- Participants at Modified High Risk for Recurrence: Participants diagnosed with locoregional RCC who underwent nephrectomy at Duke from 01 April 2014 to 31 December 2019, at modified high risk for recurrence were included. Participants at modified high risk were those who had a T stage of 3a or higher combined with a tumor grade of 2 or higher, regional lymph-node metastasis, or both.
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 119
Participants | 88

5. Primary Outcome: Number of Participants Classified According to Type of Referring Provider for Oncologic/RCC Related Care Referrals: Modified High Risk Sub-group
Description: Number of participants according to the type of provider who referred for oncologic or RCC related care after nephrectomy were recorded and reported. Type of providers included urologist, primary care, and other. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: Post-nephrectomy approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who were referred for oncologic/RCC-related care.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 31
Participants
  Urologist | 31
  Primary Care | 0
  Other | 0

6. Primary Outcome: Number of Participants Classified According to Type of Provider Referred to for Oncologic/RCC Related Care Referrals: Modified High Risk Sub-group
Description: Number of participants according to the type of provider referred to, for oncologic/RCC related care after nephrectomy were recorded and reported. Type of providers to whom participants were referred included medical oncologist, radiation oncologist, urologist, interventional radiologist, and medical geneticist. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: Post-nephrectomy approximately during 5 years (data observed during 9 months of retrospective study)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 31
Participants
  Medical Oncologist | 29
  Radiation Oncologist | 0
  Urologist | 0
  Interventional Radiology | 1
  Medical Geneticist | 1

7. Primary Outcome: Number of Participants Classified According to Reasons for Oncologic/RCC Related Care Referrals: Modified High Risk Sub-group
Description: Number of participants according to reasons for being referred to oncologic or RCC related care after nephrectomy were recorded and reported. Reasons included discussion of adjuvant systemic therapy (AST) options, other discussion of management options, and other. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: Post-nephrectomy approximately during 5 years (data observed during 9 months of retrospective study)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 31
Participants
  Discussion of AST Options | 25
  Other Discussion Management Options | 2
  Other | 4

8. Primary Outcome: Time to Any Referral for Oncologic/Renal Cell Carcinoma (RCC) Related Care: Modified High Risk Sub-group
Description: After nephrectomy, time (in days) to any referral for oncologic or RCC related care was recorded and reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: Post-nephrectomy approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who were referred for oncologic/RCC-related care and were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 27
days | 50.00 [16.00 to 812.00]

9. Primary Outcome: Time From Nephrectomy to Subsequent Surgery: Modified High Risk Sub-group
Description: Time from nephrectomy (in months) up to the subsequent surgery was recorded and reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: From nephrectomy up to the subsequent surgery, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who had any subsequent surgery after nephrectomy.
Measure: Median (Full Range); unit: months
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 5
months | 11.90 [3.21 to 22.02]

10. Primary Outcome: Number of Participants Classified According to Type of Subsequent Surgery: Modified High Risk Sub-group
Description: Number of participants according to the type of subsequent surgery after nephrectomy were reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 5
Participants
  Radical Nephrectomy | 1
  Partial Nephrectomy | 0
  Other | 4

11. Primary Outcome: Time From Nephrectomy to Receipt of First-line Adjuvant Systemic Therapy (AST): Modified High Risk Sub-group
Description: Time from nephrectomy up to the first-line AST was recorded and reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: From nephrectomy up to the first-line AST, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who received first-line AST after nephrectomy.
Measure: Median (Full Range); unit: days
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 3
days | 82.00 [76.00 to 117.00]

12. Primary Outcome: Number of Participants Classified According to Type of Systemic Agents Received as First-line AST: Modified High Risk Sub-group
Description: Number of participants according to type of systemic agents received as first-line AST were recorded and reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 3
Participants
  Sunitinib | 1
  Clinical Trial - Agent Not Specified | 2

13. Primary Outcome: Mean of Starting Dose of First-line AST Received: Modified High Risk Sub-group
Description: Mean of starting dose of first-line AST received after nephrectomy was reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: as for outcome 11
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who received first-line AST after nephrectomy and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 2
milligram | 125.00 (106.07)

14. Primary Outcome: Number of Participants Who Were Treated With First-line AST as Part of a Clinical Trial in the Adjuvant Setting: Modified High Risk Sub-group
Description: In this outcome measure number of participants who were treated with first-line AST after nephrectomy as a part of clinical trial in adjuvant setting were reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 3
Participants | 2

15. Primary Outcome: Number of Participants Classified According to First-line AST Discontinuation Reasons: Modified High Risk Sub-group
Description: In this outcome measure number of participants were classified according to reason for discontinuation of treatment with first-line AST after nephrectomy. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 2
Participants
  Adverse Event | 1
  Disease Progression | 1

16. Primary Outcome: RCC Related Follow-up Duration After Nephrectomy: Modified High Risk Sub-group
Description: RCC related follow-up duration after nephrectomy was reported. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: From nephrectomy up to the follow-up, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who were followed up related to RCC after nephrectomy.
Measure: Median (Full Range); unit: years
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 107
years | 1.57 [0.04 to 4.85]

17. Primary Outcome: Number of Participants Who Died: Modified High Risk Sub-group
Description: Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: From nephrectomy up to death by any cause, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 118
Participants | 15

18. Primary Outcome: Number of Participants Classified According to Type of Disease Recurrence: Modified High Risk Sub-group
Description: Number of participants according to the type of disease recurrence are reported. Type of disease recurrence were locoregional and distant. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: From nephrectomy up to disease recurrence, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who had RCC recurrence after nephrectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 42
Participants
  Locoregional | 4
  Distant | 38

19. Primary Outcome: Time From Nephrectomy to Recurrence: Modified High Risk Sub-group
Description: Time from nephrectomy to recurrence (in months) was defined as the time from nephrectomy to the high risk of RCC recurrence or end of participant record or receipt of systemic therapy or death due to any cause. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: as for outcome 18
Population: Analysis population included participants who were at modified high risk of recurrence. Here "Overall Number of Participants Analyzed" signifies participants who had RCC recurrence after nephrectomy and were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 40
months | 5.72 [1.02 to 46.12]

20. Other Pre Specified Outcome: Disease Free Survival (DFS): Modified High Risk Sub-group
Description: DFS was defined as the time interval (in months) from date of nephrectomy to earliest documentation of high-risk of RCC recurrence or death. Data for this outcome measure was planned to be collected and analyzed in modified high risk sub-group.
Time Frame: From nephrectomy up to earliest documentation of high-risk of recurrence or death, approximately during 5 years (data observed during 9 months of retrospective study)
Population: Analysis population included participants who were at modified high risk of recurrence.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants at Modified High Risk for Recurrence
Number analyzed (Participants) | 136
months | NA [40.60 to NA] — Median and upper limit of CI was not estimable due to low number of participants who had event.

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not collected during the study
Description: Due to non-interventional nature of the study, safety data was not collected.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT04309617/Prot_SAP_000.pdf